CLINICAL TRIAL: NCT04146870
Title: A Survey of Nutritional Status of Patients After Hematopoietic Stem Cell Transplantation
Brief Title: Nutritional Status of Patients After Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Associate Professor, The First Affiliated Hospital of Soochow University
Other Study IDs: SZnutri01
Record Dates: First submitted 2019-10-14; First posted 2019-10-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Nutrition; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: not have — not have

SUMMARY:
The main objectives of this study were :(1) to comprehensively and systematically evaluate the nutritional status of patients after hematopoietic stem cell transplantation. (2) to explore the effect of nutritional factors on the prognosis of patients treated by hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This study is devised to investigate nutritional status in patients who have undergone hematopoietic stem cell transplantation in the First Affiliated Hospital of Soochow University. Evaluation time points include the day before receiving conditioning regimen, post-transplantation 180 days, the nutritional status of patients were systematically evaluated from the aspects of food intake, physical activity level, body composition, blood biochemistry, etc. Also, the effect of nutritional factors on prognosis of hematopoietic stem cell transplantaion patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo hematopoietic stem cell transplantation in the First Affiliated Hospital of Soochow University.
* Having a life expectancy of more than 3 months

Exclusion Criteria:

* Not willing to participate in the investigation
* Age less than 15 years old or more than 80 years old

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received hematopoietic stem cell transplantation in the First Affiliated Hospital of Soochow University
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline fat free mass at 6 months | 6 months
  Body composition analyzer INBO DY S10 (bioelectrical impedance method) is used to analyze the content of fat free mass（ kilograms）
Change from Baseline fat mass at 6 months | 6 months
  Body composition analyzer INBODY S10 (bioelectrical impedance method) is used to analyze the content of fat mass（ kilograms）
Change from Baseline food intake at 6 months | 6 months
  24-hour dietary record and semi-quantitative food frequency questionnaire are used to evaluate the eating condition of patients
Change from Baseline albumin level in blood at 6 months | 6 months
  The content of albumin in blood is determined.

SECONDARY OUTCOMES:
Overall survial | 3 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive
Event free survival | 3 years
  It is measured from the date of entry into this trial to the date of relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of suzhou university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided